CLINICAL TRIAL: NCT04022850
Title: De-implementation of Low-value Pharmacological Prescriptions
Acronym: De-imFAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Health Department of the Basque Government (Unknown); Carlos III Health Institute (Other Government); European Union (Other)
Responsible Party: Principal Investigator, Alvaro Sanchez Perez, Research Technician, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2018111085; 2021111024 (Other Grant/Funding Number: Health Department of the Basque Government); PI21/00025 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII) and European Union); RD16/0007/0002 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII) and European Union); RD21/0016/0003 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII) and European Union)
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-02

CONDITIONS: Inappropriate Prescribing; Implementation Science; Behavioral Sciences

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-reflective decision assistance strategy (Active Comparator): The decision support tools integrated in the electronic health record (EHR) for the non-reflective decision assistance strategy will be applied to all FPs from the 13 Integrated Healthcare Organizations (IHOs) of Osakidetza- Basque Health Service
  Interventions: Behavioral: A non-reflective decision assistance strategy
- Reflective and non-reflective decision information strategy in addition to the previous arm (Experimental): At least 58 FPs from two IHOs (Barakaldo-Sestao and Ezkerraldea-Enkarterri-Cruces) will be randomly assigned to this experimental arm (decision assistance strategy + decision information strategy)
  Interventions: Behavioral: A non-reflective decision assistance strategy; Behavioral: A both reflective and non-reflective decision information strategy
- A reflective decision structure strategy in addition to the previous arm (Experimental): At least other 58 FPs from two IHOs (Barakaldo-Sestao and Ezkerraldea-Enkarterri-Cruces) will be randomly assigned to this experimental arm (decision assistance strategy + decision information strategy + decision structure strategy)
  Interventions: Behavioral: A non-reflective decision assistance strategy; Behavioral: A both reflective and non-reflective decision information strategy; Behavioral: A reflective decision structure strategy

INTERVENTIONS:
Behavioral: A non-reflective decision assistance strategy — A strategy based on providing evidence-based information communication technology tools to help and guide decision-making: pop-up reminders and alerts with associated messages incorporated into the REGICOR CVR calculator in OSABIDE (Osakidetza's EHR system) and within the prescription pathway in PRESBIDE (the electronic drug prescribing component).
Behavioral: A both reflective and non-reflective decision information strategy — This strategy consists of a corporate campaign entitled "Stopping Low-Value Prescribing" run by the organization (Osakidetza- Basque Health Service) that provides FPs with the evidence-based Clinical Practice Guidelines for the primary prevention of CVD in low-risk patients.
  Arms: A reflective decision structure strategy in addition to the previous arm; Reflective and non-reflective decision information strategy in addition to the previous arm
Behavioral: A reflective decision structure strategy — The strategy involves the sending of regular audit/feedback reports with practice- and organizational-level performance indicators regarding PIP of statins and healthy lifestyle promotion to prompt reflection about their own care practice, provided along with intention formation and goal-setting-focused messages.
  Arms: A reflective decision structure strategy in addition to the previous arm

SUMMARY:
The De-imFAR study is a two phase study that aims to carry out and test a structured, evidence-based and theory informed process involving the main stakeholders (managers, professionals, patients and researches) for the design, deployment, and evaluation of targeted de-implementation strategies for reducing potentially inappropriate prescribing (PIP). Specifically, the targeted low-value practice of the DE-imFAR study is the pharmacological prescription of statins in the primary prevention of cardiovascular disease (CVD) in low-risk patients. In order to prevent CVD, one of the leading causes of morbidity and death worldwide, there is general agreement on the indication of lipid-lowering treatment, mainly with statins, in patients with a cardiovascular risk (CVR) measurement greater than 10% over 10 years or in secondary prevention. Whereas, for primary prevention in patients with low CVR (<10%), preventive activities should be focused on the promotion of healthy lifestyles through optimizing diet, increasing physical activity, and stopping smoking.

Aims

1. Phase I: To design and model in a collegiate way among the agents involved (professionals, patients, managers and researchers) de-implementation strategies to favour the reduction and / or abandonment of low-value prescription of lipid-lowering drugs in primary prevention of cardiovascular disease. This strategy will be designed using systematic, comprehensive frameworks based on theory and evidence for the design of implementation strategies - the Theoretical Domains Framework (TDF) and the Behavior Change Wheel (BCW), focused on addressing the main determinants (barriers and facilitators) of clinical practice of primary prevention of CVD and adapted to the specific context of primary care in Osakidetza-Basque Health System
2. Phase II: To evaluate the effectiveness and feasibility of several de-implementation strategies derived from the systematic process of identification of determinants and mapping of adapted intervention strategies with the TDF/BCW frameworks: a strategy based on providing evidence-based information communication technology tools to help and guide decision-making (a non-reflective decision assistance strategy); a decision information strategy based on the dissemination of the evidence concerning CVD primary prevention framed in a corporate campaign encouraging family physicians to move away from PIP (a both reflective and non-reflective decision information strategy) ; and a reflective decision structure strategy encouraging reflection on actual performance based on an audit/feedback system (A reflective decision structure strategy).

Hypothesis Professionals exposed to the de-implementation strategies derived from the systematic process of identification of determinants and mapping of adapted intervention strategies with the TDF/BCW frameworks, will be effective in reducing and/or abandoning the prescription of statins in primary prevention of CVD. Among the evaluated de-implementation strategies, those that encourage self-reflection on actual performance will obtain the largest effects as compared to non-reflective strategies.

Design Phase I formative research to design and model de-implementation strategies and Phase II effectiveness and feasibility evaluation through a cluster randomized implementation trial with an additional control group. Phase I formative research will include the following actions: Cross-sectional observational study of low value pharmacological prescription in the primary prevention of CVD; Literature review on the determinants of low value pharmacological prescription behaviour and effective intervention strategies; Qualitative study on the determinants of low value pharmacological prescription in primary prevention of CVD; Collegiate mapping of the de-implementation strategies; Selection of de-implementation strategies based in perceived effectiveness and feasibility. During Phase II, the evaluation of several de-implementation strategies produced through the phase I formative evaluation will be conducted. A mixed method evaluation will be used: quantitative for assessing the implementation results at the professional level and qualitative for assessing the feasibility and perceived impact of the de-implementation strategies from the family physicians' (FPs) perspective and the experience and satisfaction of patients concerning the clinical care received.

ELIGIBILITY:
Eligibility for professionals:

* FPs belonging to any of the 13 Integrated Healthcare Organizations of Osakidetza
* Non-zero annual incidence rate of PIP of statins at baseline (2021)
* A minimum cluster size of n ≥10 patients

Eligibility for patients:

* 40- to 74-year-old men and 45- to 74-year-old women
* No history of statin use
* LDL cholesterol levels between 70 and 189 mg/dL and/or TC between 200 and 289 mg/dL
* Without ischemic heart disease/CVD
* Estimated CVR REGICOR <7.5%
* Attend at least one appointment at the participating FPs' practices during the study period from May 2022 to May 2023, and followed until May 2024

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
De-implementation strategies effectiveness: incidence of the PIP of statins | from baseline to 12 months and 24 months
  Change in the incidence of the PIP of statins recorded in the EHR in the target population.
De-implementation strategies effectiveness: incidence of the provision of advice regarding healthy lifestyles promotion activities | from baseline to 12 months and 24 months
  Change in the incidence of the provision of advice regarding healthy lifestyles promotion activities recorded in the EHR in the target population.

SECONDARY OUTCOMES:
Reach of recommendations for CVD primary prevention | 12 months
  Absolute number and percentage of patients in the target population who received the recommended CVD primary prevention clinical intervention.
De-implementation strategies secondary effectiveness: incidence of CVR (REGICOR) | from baseline to 12 months
  Change in the incidence of CVR (REGICOR) recorded in the EHR in the target population.
FP's adoption: degree to which the recommended CVD primary prevention clinical intervention is adopted by the FPs | 12 months
  Percentage of FPs who reduce PIP of statins and/or increase health promotion activities recorded in the EHR in the target population.
Strategies implementation fidelity | 12 months
  Process indicators of the delivery of and exposure to the de-implementation strategies (percentage of FPs exposed to the strategies compared)

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Bizkaia, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared that underlie results reported in the publication, after deidentification
Supporting Information: Study Protocol
Time Frame: Starting 6 months after the publication of results
Access Criteria: Since data supporting the present study will mostly concern routine data retrieved from the electronic health record of the Basque Health Service-Osakidetza, it will be only shared on justified request to the study guarantors (proposals should be directed to the Responsible Party). It will only be shared with researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Derived] Sanchez A, Pijoan JI, Sainz de Rozas R, Lekue I, San Vicente R, Quindimil JA, Rotaeche R, Etxeberria A, Mozo C, Martinez-Cengotitabengoa M, Monge M, Gomez-Ramirez C, Samper R, Ogueta Lana M, Celorrio S, Merino-Inda N, Llarena M, Gonzalez Saenz de Tejada M, Garcia-Alvarez A, Grandes G. De-imFAR phase II project: a study protocol for a cluster randomised implementation trial to evaluate the effectiveness of de-implementation strategies to reduce low-value statin prescribing in the primary prevention of cardiovascular disease. BMJ Open. 2024 Apr 17;14(4):e078692. doi: 10.1136/bmjopen-2023-078692. PMID 38631840
- [Derived] Sanchez A, Elizondo-Alzola U, Pijoan JI, Mediavilla MM, Pablo S, Sainz de Rozas R, Lekue I, Gonzalez-Larragan S, Llarena M, Larranaga O, Helfrich CD, Grandes G. Applying the behavior change wheel to design de-implementation strategies to reduce low-value statin prescription in primary prevention of cardiovascular disease in primary care. Front Med (Lausanne). 2022 Oct 13;9:967887. doi: 10.3389/fmed.2022.967887. eCollection 2022. PMID 36314033
- [Derived] Sanchez A, Pijoan JI, Pablo S, Mediavilla M, de Rozas RS, Lekue I, Gonzalez-Larragan S, Lantaron G, Argote J, Garcia-Alvarez A, Latorre PM, Helfrich CD, Grandes G. Addressing low-value pharmacological prescribing in primary prevention of CVD through a structured evidence-based and theory-informed process for the design and testing of de-implementation strategies: the DE-imFAR study. Implement Sci. 2020 Jan 22;15(1):8. doi: 10.1186/s13012-020-0966-3. PMID 31969175